CLINICAL TRIAL: NCT00006105
Title: Phase II Trial of Adjuvant Gemcitabine Plus Cisplatin With Amifostine Cytoprotection in Patients With Locally Advanced Bladder Cancer
Brief Title: Gemcitabine, Cisplatin, and Amifostine Following Surgery in Treating Patients With Locally Advanced Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9193; UCCRC-9193; UCCRC-CTRC-9806; NCI-G00-1831
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Bladder Cancer; Drug/Agent Toxicity by Tissue/Organ
Keywords: stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer; drug/agent toxicity by tissue/organ
MeSH Terms: conditions — Urinary Bladder Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — Amifostine; Cisplatin; Gemcitabine; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Administration of Cisplatin, Gemcitabine, and Amifostine (Experimental): Subjects receive the study drug combination in 29-day cycles. Gemcitabine (1000 mg/m2) is given by IV infusion on Days 1, 8, and 15 of each cycle. Cisplatin (70 mg/m2) is given by IV infusion on Day 1 of each cycle. Immediately prior to each cisplatin infusion amifostine (910 mg/m2) will be given by IV infusion.
  Interventions: Drug: amifostine trihydrate; Drug: cisplatin; Drug: gemcitabine hydrochloride; Procedure: adjuvant therapy

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Drug: gemcitabine hydrochloride
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine, cisplatin, and amifostine following surgery in treating patients who have locally advanced bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of adjuvant gemcitabine and cisplatin with amifostine cytoprotection in patients with completely resected locally advanced bladder cancer.
* Compare recurrence rate in these patients when treated with this regimen to historical control patients who had a cystectomy performed by the same surgeon.

OUTLINE: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15, and cisplatin IV over 60 minutes and amifostine IV over 15 minutes on day 1. Treatment continues every 28 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 19-42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Completely resected locally advanced bladder cancer

  * T2-4, N0-2
* Post radical cystectomy with no gross residual disease
* No evidence of metastases by CT of chest, abdomen, and pelvis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL (transfusion allowed)

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST and ALT no greater than 3 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 50 mL/min

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study participation
* No active infection
* No serious concurrent systemic disorders that would preclude study participation
* No metastatic cancer in past 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except contraceptives and replacement steroids

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 but no more than 8 weeks since radical cystectomy

Other:

* No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2000-06; Primary Completion 2004-11 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Side effects of cisplatin/gemcitabine in combination with amifostine | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Walter M. Stadler, MD, FACP, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States